CLINICAL TRIAL: NCT03144479
Title: A New Technique to Assess the Correct Positioning of a Right-sided Double-lumen Tube Without Fiberoptic Bronchoscopy
Brief Title: New Technique to Assess Correct Positioning of the Right-sided Double Lumen Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016/29dec/565
Record Dates: First submitted 2017-03-29; First posted 2017-05-08 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Anesthesia; Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positioning of right-sided double lumen tube with fluoroscopy (Experimental): positioning of the right-sided double lumen tube with a wire guide and fluoroscopy
  Interventions: Procedure: right-sided double lumen tube
- Positioning of right-sided double lumen tube with fibroscope (Experimental): positioning of the right sided double lumen tube in the same patient but with a fibroscope
  Interventions: Procedure: right-sided double lumen tube

INTERVENTIONS:
Procedure: right-sided double lumen tube — Verification of a new technique to assess the correct positioning of a right-sided double-lumen tube for left thoracic surgeries, using a central venous catheter wire guide and a radioscopy
  Other Names: Device intervention : central venous catheter wire guide and radioscopy

SUMMARY:
A technique not yet described in the literature and allowing anesthesiologists who do not regularly practice fibroscopy or who do not routinely have this type of apparatus for their procedures, to install straight double-lumen tubes without compromising the ventilation of the patient. The aim is to introduce a central venous catheter wire guide into the bronchial arm of the right double-lumen tube and insert it into the right upper lobe bronchus orifice under fluoroscopic control. Then, to validate the new technique, we will carry out a fibroscopic control.

DETAILED DESCRIPTION:
Right-sided double lumen tube (Mallinckrodt - Endobronchial tube) is introduced into the glottis via direct laryngoscopy. After the endotracheal lumen tube has passed the vocal cords, the stylet is removed, and the tube is rotated 90° toward the right and advanced slightly until resistance is encountered. Auscultation is then performed to check the proper side the endobronchial tube was inserted to.

Then, the anatomy of the carina and the origins of the right and left upper bronchus are identified with the video-bronchoscopy.

After a mild plication of the distal extremity of an adult central venous catheter wire guide (0.53mm diameter, 45cm length, one straight soft tip on one end and one "J" tip on other), the J-shaped extremity of this guide is introduced through the endobronchial lumen under direct video-bronchoscope. The wire guide is then slowly removed in order that proper alignment between the wire extremity and the right upper lobe occurs. The wire is removed again until its J-shaped extremity appears through the right-upper lobe ventilation orifice. In order to align the orifice of the tube with the upper lobe bronchus, a rotational movement of the double-lumen tube may be necessary. When the location of the orifice of the right upper lobe is identified, the guide is moved forward through the orifice into the upper lobe bronchus.

Once satisfactory initial placement is achieved, the bronchial cuff is left inflated, the wire guide of the central venous catheter is kept in place in the upper lobe bronchus, and the patient is turned to the right lateral decubitus position. The proper positioning of the tube is once again checked by another video-bronchoscopy.

To confirm the exact placement of the tube, a fiberoptic bronchoscopy is performed through the endobronchial lumen to find the right upper lobe ventilation orifice and confirm alignment. Then, it is placed distally to the endobronchial lumen to confirm a clear view showing the bronchus intermedius.

After passing the fiberoptic bronchoscope through the tracheal lumen, the blue bronchial cuff is visualized at the origin of the right main stem bronchus below the level of the carina.

ELIGIBILITY:
Inclusion Criteria:

* all patients > 18 years old who have to undergo a left thoracic surgery with a one lung ventilation technique

Exclusion Criteria:

* emergency surgical procedures, patients with predictable difficulties of insertion of a double-lumen endotracheal tube, hemodynamically unstable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of the distance between the lateral orifice of the tube and the orifice of the right upper lobe bronchus | 20 minutes
  Fibroscopic measurement to assess the correct positioning of the right-sided double lumen tube with the wire guide and the fluoroscopy

SECONDARY OUTCOMES:
Total time spent to correctly position the right-sided double lumen tube | 20 minutes
  If the technique with the wire guide and the fluoroscopy, takes more than 20 minutes to be achieved, it is considered as failed.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Watremez, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campos JH, Massa FC, Kernstine KH. The incidence of right upper-lobe collapse when comparing a right-sided double-lumen tube versus a modified left double-lumen tube for left-sided thoracic surgery. Anesth Analg. 2000 Mar;90(3):535-40. doi: 10.1097/00000539-200003000-00007. PMID 10702432
- [Result] de Bellis M, Accardo R, Di Maio M, La Manna C, Rossi GB, Pace MC, Romano V, Rocco G. Is flexible bronchoscopy necessary to confirm the position of double-lumen tubes before thoracic surgery? Eur J Cardiothorac Surg. 2011 Oct;40(4):912-6. doi: 10.1016/j.ejcts.2011.01.070. Epub 2011 Jul 29. PMID 21802958